CLINICAL TRIAL: NCT01396421
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Three Fixed Doses of OPC-34712 in the Treatment of Adults With Acute Schizophrenia
Brief Title: Study of the Effectiveness of Three Different Doses of OPC-34712 in the Treatment of Adults With Acute Schizophrenia
Acronym: VECTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-10-231
Record Dates: First submitted 2011-07-11; First posted 2011-07-18 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-09

CONDITIONS: Acute Schizophrenia
MeSH Terms: interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- OPC-34712 [Brexpiprazole] High Dose (Experimental): Higher Dose, tablet, once daily, for six weeks
  Interventions: Drug: OPC-34712 [Brexpiprazole] High Dose
- OPC-34712 [Brexpiprazole] Middle Dose (Experimental): Middle Dose, tablet, once daily, for six weeks
  Interventions: Drug: Experimental: OPC-34712 [Brexpiprazole] Middle Dose
- OPC-34712 [Brexpiprazole] Low Dose (Experimental): Lower Dose, tablet, once daily, for six weeks
  Interventions: Drug: Experimental: OPC-34712 [Brexpiprazole] Low Dose
- Placebo (Placebo Comparator): Placebo, once daily, for six weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-34712 [Brexpiprazole] High Dose — Higher dose, tablet, once daily, for six weeks
  Arms: OPC-34712 [Brexpiprazole] High Dose
Drug: Experimental: OPC-34712 [Brexpiprazole] Middle Dose — Middle dose, tablet, once daily, for six weeks
  Arms: OPC-34712 [Brexpiprazole] Middle Dose
Drug: Experimental: OPC-34712 [Brexpiprazole] Low Dose — Lower dose, tablet, once daily, for six weeks
  Arms: OPC-34712 [Brexpiprazole] Low Dose
Drug: Placebo — Placebo, once daily, for six weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effectiveness, safety and tolerability of three different doses of OPC-34712 with placebo in the treatment of acute schizophrenia in adults.

DETAILED DESCRIPTION:
Schizophrenia is a severely debilitating mental illness that affects approximately 1% of the world population. Hallucinations and delusions are the most striking characteristic positive symptoms of schizophrenia; however, more subtle negative symptoms (eg, social withdrawal and lack of emotion, energy, and motivation) may also be present. The first antipsychotics developed for the treatment of schizophrenia were effective against positive symptoms, but showed little efficacy for negative symptoms and were also associated with a high incidence of side effects. Second generation antipsychotics, represent a significant advancement in the treatment of psychotic disorders because they are effective and at the same time exhibit fewer side effects than first generation antipsychotics. Although generally safer than first generation antipsychotics, the second-generation antipsychotics are not devoid of undesirable side effects such as Hyperprolactinemia and weight gain. In addition, the safety of these drugs vary considerably.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 65 years of age, with a diagnosis of schizophrenia, as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria
2. Subjects who have been recently hospitalized or who would benefit from hospitalization for an acute relapse of schizophrenia
3. Subjects experiencing an acute exacerbation of psychotic symptoms
4. Other protocol specific inclusion criteria may apply

Exclusion Criteria:

1. Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug
2. Subjects with a current DSM-IV-TR Axis I diagnosis of:

   * Schizoaffective disorder
   * Major depressive disorder (MDD)
   * Bipolar disorder
   * Delirium, dementia, amnestic or other cognitive disorder
   * Borderline, paranoid, histrionic, schizotypal, schizoid or antisocial personality disorder
3. Subjects presenting with a first episode of schizophrenia
4. Other protocol specific exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Skuban, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (49):
- United States (15):
  - Little Rock, Arkansas
  - Garden Grove, California
  - Glendale, California
  - Oakland, California
  - Oceanside, California
  - San Diego, California
  - Bradenton, Florida
  - Miami Springs, Florida
  - Orlando, Florida
  - Fresh Meadows, New York
  - Jamaica, New York
  - Dayton, Ohio
  - Charleston, South Carolina
  - Austin, Texas
  - Kirkland, Washington
- Canada (2):
  - Burlington, Ontario
  - Chatham, Ontario
- Japan (5):
  - Fujisawa-shi, Kanagawa
  - Kunigami-gun, Okinawa
  - Sakai-shi, Osaka
  - Setagaya-ku, Tokyo-To
  - Kumamoto
- Latvia (5):
  - Daugavpils
  - Jelgava
  - Liepāja
  - Riga
  - Strenči
- Poland (3):
  - Choroszcz
  - Gdansk
  - Lodz
- Romania (6):
  - Arad
  - Bucharest
  - Cluj-Napoca
  - Focşani
  - Piteşti
  - Târgovişte
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Novi Sad
- South Korea (2):
  - Incheon
  - Seoul
- Ukraine (8):
  - Chernihiv
  - Dnipropetrovsk
  - Hlevakha
  - Kherson, Vil. Stepanivka
  - Kyiv
  - Lviv
  - Simferopol
  - Vinnytsia

REFERENCES:
- [Derived] Ismail Z, Kapadia S, Palma AM, Yildirim M, Farovik A. Brexpiprazole for anxiety symptoms in schizophrenia: a pooled analysis of short- and long-term trials. Curr Med Res Opin. 2025 Aug;41(8):1535-1548. doi: 10.1080/03007995.2025.2552286. Epub 2025 Sep 11. PMID 40859756
- [Derived] Ismail Z, Meehan SR, Farovik A, Kapadia S, Palma AM, Zhang Z, McIntyre RS. Effects of brexpiprazole on patient life engagement in schizophrenia: post hoc analysis of Positive and Negative Syndrome Scale data. Curr Med Res Opin. 2025 Jan;41(1):145-153. doi: 10.1080/03007995.2024.2440059. Epub 2025 Jan 3. PMID 39749727
- [Derived] Correll CU, He Y, Therrien F, MacKenzie E, Meehan SR, Weiss C, Hefting N, Hobart M. Effects of Brexpiprazole on Functioning in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. J Clin Psychiatry. 2022 Mar 1;83(2):20m13793. doi: 10.4088/JCP.20m13793. PMID 35235720
- [Derived] Marder SR, Meehan SR, Weiss C, Chen D, Hobart M, Hefting N. Effects of Brexpiprazole Across Symptom Domains in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. Schizophr Bull Open. 2021 May 1;2(1):sgab014. doi: 10.1093/schizbullopen/sgab014. eCollection 2021 Jan. PMID 34901863
- [Derived] Newcomer JW, Eriksson H, Zhang P, Weiller E, Weiss C. Changes in metabolic parameters and body weight in brexpiprazole-treated patients with acute schizophrenia: pooled analyses of phase 3 clinical studies. Curr Med Res Opin. 2018 Dec;34(12):2197-2205. doi: 10.1080/03007995.2018.1498779. Epub 2018 Jul 27. PMID 29985680
- [Derived] Kane JM, Skuban A, Hobart M, Ouyang J, Weiller E, Weiss C, Correll CU. Overview of short- and long-term tolerability and safety of brexpiprazole in patients with schizophrenia. Schizophr Res. 2016 Jul;174(1-3):93-98. doi: 10.1016/j.schres.2016.04.013. Epub 2016 May 14. PMID 27188270
- [Derived] Correll CU, Skuban A, Ouyang J, Hobart M, Pfister S, McQuade RD, Nyilas M, Carson WH, Sanchez R, Eriksson H. Efficacy and Safety of Brexpiprazole for the Treatment of Acute Schizophrenia: A 6-Week Randomized, Double-Blind, Placebo-Controlled Trial. Am J Psychiatry. 2015 Sep 1;172(9):870-80. doi: 10.1176/appi.ajp.2015.14101275. Epub 2015 Apr 16. PMID 25882325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 636 participants from 65 trial sites in 10 countries.
Pre-assignment Details: Adults with schizophrenia as defined by Diagnostic and Statistical Manual of Mental Health Disorders 4th Edition Text Revision criteria and confirmed by the Mini International Neuropsychiatric Interview for schizophrenia and psychotic disorders studies.
Groups:
- Brexpiprazole 4 mg: Brexpiprazole 4 milligram (mg) tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 1-week period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2).
- Brexpiprazole 2mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 5 day period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose by Day 5.
- Brexpiprazole 0.25mg: Brexpiprazole 0.25mg tablet once daily for 6 weeks.
- Placebo: Placebo tablet once daily for 6 weeks.
Period: Overall Study
Arm/Group | Brexpiprazole 4 mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Started | 180 | 182 | 90 | 184
Completed | 121 | 124 | 56 | 109
Not Completed | 59 | 58 | 34 | 75
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Adverse Event | 17 | 15 | 12 | 32
Not completed — Participant Met Withdrawal Criteria | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 31 | 24 | 13 | 21
Not completed — Protocol Deviation | 2 | 1 | 1 | 0
Not completed — Lack of Efficacy | 7 | 17 | 7 | 18

BASELINE CHARACTERISTICS:
Groups:
- Brexpiprazole 4mg: Brexpiprazole 4mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 1-week period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2).
- Brexpiprazole 0.25 mg: Brexpiprazole 0.25mg tablet once daily for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25 mg | Placebo | Total
Number analyzed (Participants) | 180 | 182 | 90 | 184 | 636
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (11.0) | 39.6 (10.2) | 40.5 (11.4) | 39.7 (10.8) | 40.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 71 | 29 | 66 | 235
  Male | 111 | 111 | 61 | 118 | 401

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 6 Positive and Negative Syndrome Scale (PANSS) Total Score.
Description: The PANSS consists of 3 subscales (positive subscale, negative subscale and general psychology subscale) containing a total of 30 symptom constructs and was administered using the Structured Clinical Interview (SCI)-PANSS. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline to Week 6
Population: Efficacy: consists of all participants who received at least one dose of study medication and have baseline and at least one post-baseline efficacy evaluation. At Week 6, 134, 132, 62 and 124 participants in the Brex 4mg, Brex 2mg, Brex 0.25 mg and placebo group, respectively had data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole 4mg: Brexpiprazole 4mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 1-week period beginning at the randomization (Day 1),and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2).
- Brexpiprazole 2 mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 5 day period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose by Day 5.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2 mg | Brexpiprazole 0.25 mg | Placebo
Number analyzed (Participants) | 134 | 132 | 62 | 124
Units on a scale | -19.65 (1.54) | -20.73 (1.55) | -14.90 (2.23) | -12.01 (1.60)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Brexpiprazole 2 mg vs Placebo; Difference between average effect of brexpiprazole 2 and 4 mg/day and placebo was tested first at alpha level of 0.05. If statistically significant, then comparisons for each group (brexpiprazole 2 and 4 mg/day) versus placebo were performed; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Primary analysis was performed by fitting a Mixed Model Repeated Measures (MMRM) which included fixed class effect terms for treatment, trial site, visit week, and an interaction term of treatment by visit week; MMRM with fixed effect of treatment, clinical center, visit, treatment visit interaction, baseline value, baseline visit interaction as covariates; Treatment difference = -8.18, 95% CI 2-sided [-12.0 to -4.40]
Statistical Analysis 2: Comparison: Brexpiprazole 4mg vs Placebo; Sample size was determined to achieve 90% power at alpha level of 0.025 (two-sided) to a detect treatment difference of -7.5 points in change from baseline in PANSS Total Score at Week 6 (last observation carried forward) between a brexpiprazole treatment of 4 mg/day (or 2 mg/day) and placebo using a two-sided z-test; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Treatment difference = -7.64, 95% CI 2-sided [-12.0 to -3.30]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Traetment difference = -8.72, 95% CI 2-sided [-13.1 to -4.37]
Statistical Analysis 4: Comparison: Brexpiprazole 0.25 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2910, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Treatment difference = -2.89, 95% CI 2-sided [-8.27 to 2.49]

2. Secondary Outcome: Mean Change From Baseline to Week 6 in Clinical Global Impression - Severity of Illness Scale (CGI-S) Score.
Description: The severity of illness was rated using the CGI-S which is the key secondary endpoint. To perform this assessment, the rater or study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0=not assessed; 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill participant.
Time Frame: Baseline to Week 6
Population: Efficacy: consists of all participants who received at least one dose of study medication and have baseline and at least one post-baseline efficacy evaluation. At Week 6, 121, 124, 56 and 109 participants in the Brex 4mg, Brex 2mg, Brex 0.25 mg and placebo group, respectively had data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole 4 mg: Brexpiprazole 4mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 1-week period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2).
Arm/Group | Brexpiprazole 4 mg | Brexpiprazole 2 mg | Brexpiprazole 0.25 mg | Placebo
Number analyzed (Participants) | 121 | 124 | 56 | 109
Units on a scale | -1.20 (0.08) | -1.15 (0.08) | -0.85 (0.12) | -0.82 (0.09)
Statistical Analysis 1: Comparison: Brexpiprazole 4 mg vs Brexpiprazole 2 mg vs Placebo; Difference between the average effect of brexpiprazole 2 and 4 mg/day and placebo was tested first at alpha level of 0.05. If statistically significant, then comparisons for each group (brexpiprazole 2 and 4 mg/day) versus placebo were performed at a significance level of 0.05; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.36, 95% CI 2-sided [-0.56 to -0.15]
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg vs Placebo; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.38, 95% CI 2-sided [-0.61 to -0.15]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg vs Placebo; Test type: Superiority or Other; p = 0.0056, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.33, 95% CI 2-sided [-0.56 to -0.10]
Statistical Analysis 4: Comparison: Brexpiprazole 0.25 mg vs Placebo; Test type: Superiority or Other; p = 0.8491, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.03, 95% CI 2-sided [-0.31 to 0.26]

3. Secondary Outcome: Mean Change From Baseline to Week 1, 2, 3, 4 and 5 Positive and Negative Syndrome Scale (PANSS) Total Score.
Description: as for outcome 1
Time Frame: Baseline to Week 1, 2, 3, 4, 5
Population: Efficacy: consists of all participants who received at least one dose of study medication and have baseline and at least one post-baseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole 2mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 5 day period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose by Day 5).
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 178 | 180 | 87 | 178
Units on a scale
  Week 1 | -4.38 (0.60) | -4.87 (0.59) | -2.52 (0.83) | -2.87 (0.60)
  Week 2 | -9.51 (0.93) | -8.86 (0.93) | -3.28 (1.32) | -5.11 (0.95)
  Week 3 | -12.78 (1.15) | -11.08 (1.16) | -5.71 (1.65) | -7.64 (1.18)
  Week 4 | -16.50 (1.32) | -14.06 (1.32) | -8.86 (1.90) | -8.89 (1.35)
  Week 5 | -18.61 (1.42) | -17.90 (1.43) | -11.87 (2.05) | -10.75 (1.47)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0644, Mixed Models Analysis — MMRM with fixed effect of treatment, (pooled) clinical center, visit, treatment visit interaction, baseline value, and baseline visit interaction as covariates; Week 1; Treatment difference = -1.50, 95% CI 2-sided [-3.09 to 0.09]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0139, Mixed Models Analysis — MMRM with fixed effect of treatment, (pooled) clinical center, visit, treatment visit interaction, baseline value, baseline visit interaction as covariates; Week 1; Treatment difference = -1.99, 95% CI 2-sided [-3.58 to -0.41]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.7231, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 1; Treatment difference = 0.35, 95% CI 2-sided [-1.61 to 2.32]
Statistical Analysis 4: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 3; Treatment difference = -5.14, 95% CI 2-sided [-8.36 to -1.93]
Statistical Analysis 5: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0045, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 2; Treatment difference = -3.75, 95% CI 2-sided [-6.33 to -1.17]
Statistical Analysis 6: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.2568, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 2; Treatment difference = 1.84, 95% CI 2-sided [-1.34 to 5.02]
Statistical Analysis 7: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 2; Treatment difference = -4.40, 95% CI 2-sided [-6.97 to -1.82]
Statistical Analysis 8: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0360, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 3; Treatment difference = -3.45, 95% CI 2-sided [-6.67 to -0.23]
Statistical Analysis 9: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.9876, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 4; Treatment difference = 0.04, 95% CI 2-sided [-4.53 to 4.60]
Statistical Analysis 10: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 4; Treatment difference = -7.61, 95% CI 2-sided [-11.3 to -3.93]
Statistical Analysis 11: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0062, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 4; Treatment difference = -5.16, 95% CI 2-sided [-8.85 to -1.47]
Statistical Analysis 12: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.3407, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 3; Treatment difference = 1.93, 95% CI 2-sided [-2.05 to 5.90]
Statistical Analysis 13: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 5; Treatment difference = -7.86, 95% CI 2-sided [-11.9 to -3.86]
Statistical Analysis 14: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 5; Treatment difference = -7.15, 95% CI 2-sided [-11.2 to -3.14]
Statistical Analysis 15: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.6570, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 5; Treatment difference = -1.12, 95% CI 2-sided [-6.07 to 3.83] — Because only the comparison of brexpiprazole 4 mg/day versus placebo met the threshold in the primary analysis, the following analysis is not part for the formal statistical testing and is descriptive only

4. Secondary Outcome: Mean Change From Baseline to Week 1, 2, 3, 4 and 5 in Clinical Global Impression - Severity of Illness Scale (CGI-S) Score.
Description: The severity of illness was rated using the CGI-S. To perform this assessment, the rater or study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0=not assessed; 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill participant.
Time Frame: Baseline to Week 1, 2, 3, 4 and 5
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 178 | 181 | 89 | 181
Units on a scale
  Week 1 | -0.16 (0.04) | -0.16 (0.04) | -0.11 (0.05) | -0.14 (0.04)
  Week 2 | -0.46 (0.05) | -0.43 (0.05) | -0.18 (0.07) | -0.30 (0.05)
  Week 3 | -0.72 (0.06) | -0.60 (0.06) | -0.33 (0.09) | -0.51 (0.07)
  Week 4 | -0.96 (0.07) | -0.73 (0.07) | -0.58 (0.11) | -0.54 (0.08)
  Week 5 | -1.08 (0.08) | -1.03 (0.08) | -0.73 (0.11) | -0.69 (0.08)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.6553, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 1; Treatment difference = -0.02, 95% CI 2-sided [-0.13 to 0.08]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.6170, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 1; Treatment difference = -0.03, 95% CI 2-sided [-0.13 to 0.08]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.6446, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 1; Treatment difference = 0.03, 95% CI 2-sided [-0.10 to 0.15]
Statistical Analysis 4: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0347, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 2; Treatment difference = -0.15, 95% CI 2-sided [-0.29 to -0.01]
Statistical Analysis 5: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0825, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Leasr squares mean = -0.12, 95% CI 2-sided [-0.27 to 0.02]
Statistical Analysis 6: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.1678, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 2; Treatment difference = 0.12, 95% CI 2-sided [-0.05 to 0.30]
Statistical Analysis 7: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0219, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 3; Treatment difference = -0.21, 95% CI 2-sided [-0.39 to -0.03]
Statistical Analysis 8: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.3275, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 3; Least squares mean = -0.09, 95% CI 2-sided [-0.27 to 0.09]
Statistical Analysis 9: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.1173, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 3; Treatment difference = 0.18, 95% CI 2-sided [-0.04 to 0.40]
Statistical Analysis 10: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 4; Treatment difference = -0.42, 95% CI 2-sided [-0.63 to -0.21]
Statistical Analysis 11: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0662, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 4; Least squares mean = -0.19, 95% CI 2-sided [-0.40 to 0.01]
Statistical Analysis 12: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.7587, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 4; Treatment difference = -0.04, 95% CI 2-sided [-0.30 to 0.22]
Statistical Analysis 13: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 5; Treatment difference = -0.39, 95% CI 2-sided [-0.61 to -0.17]
Statistical Analysis 14: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0032, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 5; Least squares mean = -0.34, 95% CI 2-sided [-0.56 to -0.11]
Statistical Analysis 15: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.7619, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 5; Treatment difference = -0.04, 95% CI 2-sided [-0.32 to 0.23]

5. Secondary Outcome: Mean Change From Baseline to Week 6 in Personal and Social Performance Scale (PSP)
Description: The PSP is a clinician-rated scale that measures personal and social functioning in 4 domains: socially useful activities (eg, work and study), personal and social relationships, self-care, and disturbing and aggressive behaviors. Impairment in each of these domains was rated as absent, mild, manifest, marked, severe, or very severe. These ratings were then converted to a total score based on a 100-point scale using algorithms to identify the appropriate 10-point interval, and the rater's judgment to determine the total score within the 10-point interval. Participants with a PSP total score of 71 to 100 were considered to have mild functional difficulty. Scores of 31 to 70 represented manifest disabilities of various degrees and ratings of 1 to 30 indicated minimal functioning that required intense support and/or supervision.
Time Frame: Baseline to Week 6
Population: Efficacy: consists of all participants who received at least one dose of study medication and have baseline and at least one post-baseline efficacy evaluation. At Week 6, 121, 122, 55 and 108 participants in the Brex 4mg, Brex 2mg, Brex 0.25 mg and placebo group, respectively had data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole 2mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a r5 day period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose by Day 5.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 122 | 55 | 108
Units on a scale | 12.72 (0.93) | 13.15 (0.93) | 11.84 (1.33) | 10.26 (0.98)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0557, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 6; Treatment difference = 2.46, 95% CI 2-sided [-0.06 to 4.98]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0250, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 6; Treatment difference = 2.89, 95% CI 2-sided [0.37 to 5.42]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.3264, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Week 6; Treatment difference = 1.58, 95% CI 2-sided [-1.58 to 4.74]

6. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Positive Subscale Score
Description: For each symptom construct of the PANSS Positive Subscale, severity was rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. The symptom constructs were as follows: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS Positive Subscale Score for each participant was calculated as the sum of the rating assigned to each of the 7 subscale items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline to Week 6
Population: Efficacy: consists of all participants who received at least one dose of study medication and have baseline and at least one post-baseline efficacy evaluation. At Week 6, 121, 123, 56 and 108 participants in the Brex 4mg, Brex 2mg, Brex 0.25 mg and placebo group, respectively had data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole 2mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 1-week period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2).
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 123 | 56 | 108
Units on a scale | -6.78 (0.51) | -6.57 (0.52) | -5.46 (0.74) | -4.35 (0.54)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -2.44, 95% CI 2-sided [-3.88 to -0.99]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -2.22, 95% CI 2-sided [-3.67 to -0.77]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.2227, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.11, 95% CI 2-sided [-2.90 to 0.68]

7. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Negative Subscale Score
Description: For each symptom construct of the PANSS Negative Subscale, severity was rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. The symptom constructs were as follows: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS Negative Subscale Score for each participant was calculated as the sum of the rating assigned to each of the 7 subscale items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 123 | 56 | 108
Units on a scale | -3.65 (0.36) | -4.02 (0.36) | -3.31 (0.53) | -2.24 (0.38)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0069, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.41, 95% CI 2-sided [-2.44 to 0.39]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Least squares mean = -1.78, 95% CI 2-sided [-2.81 to -0.76]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.0996, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatmetn difference = -1.07, 95% CI 2-sided [-2.33 to 0.20]

8. Secondary Outcome: Clinical Global Impression- Improvement Scale (CGI-I) Score at Week 6
Description: The participant's overall improvement was rated using the CGI-I. The rater or study physician rated the participant's total improvement whether or not it was due entirely to drug treatment. All responses were compared with the participant's condition at screening/baseline. Response choices were: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse.
Time Frame: Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Brexpiprazole 4mg: Brexpiprazole 4mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 1-week period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 178 | 181 | 89 | 178
Units on a scale | 2.94 (1.29) | 2.94 (1.34) | 3.37 (1.46) | 3.48 (1.47)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel — The Cochran-Mantel-Haenzel (CMH) row mean scores differ test controlling for trial center was applied to CGI-I score; Treatment difference = -0.50, 95% CI 2-sided [-0.77 to -0.22]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — The CMH row mean scores differ test controlling for trial center was applied to CGI-I score; Treatment difference = -0.54, 95% CI 2-sided [-0.82 to -0.26]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.4505, Cochran-Mantel-Haenszel — The CMH row mean scores differ test controlling for trial center was applied to CGI-I score; Treatment difference = -0.14, 95% CI 2-sided [-0.50 to 0.22]

9. Secondary Outcome: Response Rate at Week 6
Description: Response rate was defined as improvement in mean change of ≥30% from baseline in PANSS Total Score at Week 6 or CGI-I score of 1 (very much improved) or 2 (much improved) at Week 6.
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Groups:
- Brexpiprazole 2mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 5-day period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose by Day 5.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 178 | 180 | 87 | 178
Percentage of participants | 46.07 | 47.78 | 39.08 | 30.34
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0032, Cochran-Mantel-Haenszel — CMH general association test controlling for trial was applied to the analysis of response rate; Relative risk = 1.48, 95% CI 2-sided [1.14 to 1.91]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel — CMH general association test controlling for trial was applied to the analysis of response rate; Relative risk = 1.59, 95% CI 2-sided [1.23 to 2.05]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.1576, Cochran-Mantel-Haenszel — CMH general association test controlling for trial was applied to the analysis of response rate; Relative risk = 1.27, 95% CI 2-sided [0.92 to 1.76]

10. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Excited Component (PEC) Score
Description: The PEC consists of 5 PANSS items (excitement [P4], hostility [P7], tension [G4], uncooperativeness [G8], and poor impulse control [G14]). Each rated on a scale of 1 (absent) to 7 (extreme). The PEC for participants was calculated as the sum of the rating assigned to each of the 5 items, and ranged from 5 to 35 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole 2mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 5-day period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day by Day 5.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 123 | 56 | 108
Units on a scale | -2.75 (0.34) | -2.87 (0.34) | -1.99 (0.49) | -1.64 (0.36)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0246, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.10, 95% CI 2-sided [-2.06 to -0.14]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0131, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.22, 95% CI 2-sided [-2.19 to -0.26]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.5706, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -0.34, 95% CI 2-sided [-1.53 to 0.85]

11. Secondary Outcome: Discontinuation Rate for Lack of Efficacy at Week 6
Time Frame: Week 6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 178 | 180 | 87 | 178
Percentage of participants | 3.93 | 9.44 | 8.05 | 10.11
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0143, Cochran-Mantel-Haenszel; CMH general association test controlling for trial center was applied to the analysis of discontinuation rate; Relative risk = 0.39, 95% CI 2-sided [0.18 to 0.85]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.6606, Cochran-Mantel-Haenszel — CMH general association test controlling for trial center was applied to the analysis of discontinuation rate; Relative risk = 0.87, 95% CI 2-sided [0.46 to 1.65]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.5115, Cochran-Mantel-Haenszel — CMH general association test controlling for trial center was applied to the analysis of discontinuation rate; Relative risk = 0.77, 95% CI 2-sided [0.35 to 1.68]

12. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Factor Score - Positive Symptoms Score
Description: The PANSS Marder Factor score - Positive Symptoms Score consists of 8 PANSS items (delusions [P1], hallucinatory behaviour [P3], grandiosity [P5], suspiciousness [P6], stereotyped thinking [N7], somatic concern [G1], unusual thought content [G9], lack of judgment and insight [G10]. Each was rated on a scale of 1 (absent) to 7 (extreme). The PANSS Marder Factor score - Positive Symptoms Score for participants was calculated as the sum of the rating assigned to each of the 8 items, and ranged from 8 to 42 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 123 | 56 | 108
Units on a scale | -7.23 (0.51) | -7.37 (0.51) | -5.78 (0.73) | -4.89 (0.53)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -2.34, 95% CI 2-sided [-3.77 to -0.91]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -2.47, 95% CI 2-sided [-3.91 to -1.04]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.3263, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -0.89, 95% CI 2-sided [-2.66 to 0.89]

13. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Factor Score - Negative Symptoms Score
Description: The PANSS Marder Factor score - Negative Symptoms Score consists of 7 PANSS items (blunted effect [N1], emotional withdrawal [N2], poor rapport [N3], passive/apathetic social withdrawal [N4], lack of spontaneity and conversation flow [N6], motor retardation [G7], active social avoidance [G16]). The PANSS Marder Factor score - Negative Symptoms Score for participants was calculated as the sum of the rating assigned to each of the 7 items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 123 | 56 | 108
Units on a scale | -4.10 (0.37) | -4.48 (0.37) | -3.66 (0.54) | -2.80 (0.38)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0155, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.30, 95% CI 2-sided [-2.35 to -0.25]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.68, 95% CI 2-sided [-2.73 to -0.62]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.1956, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -0.86, 95% CI 2-sided [-2.17 to 0.44]

14. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Disorganised Thought Score
Description: The PANSS Marder Factor score -Disorganized Thought Score consists of 7 PANSS items (conceptual disorganization [P2], difficulty in abstract thinking [N5], mannerisms and posturing [G5], disorientation [G10], poor attention [G11], disturbance of violation [G13], preoccupation [G15]). The PANSS Marder Factor score - Disorganized Thought Score for participants was calculated as the sum of the rating assigned to each of the 7 items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 123 | 56 | 108
Units on a scale | -3.72 (0.36) | -3.94 (0.36) | -2.69 (0.52) | -1.97 (0.37)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.75, 95% CI 2-sided [-2.76 to -0.75]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.98, 95% CI 2-sided [-2.98 to -0.97]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.2572, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -0.72, 95% CI 2-sided [-1.96 to 0.52]

15. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Uncontrolled Hostility/Excitement Score
Description: The PANSS Marder Factor score - Uncontrolled Hostility/Excitement Score consists of 4 PANSS items (excitement [P4], hostility [P7], uncooperativeness [G8], poor impulse control [G14]). The PANSS Marder Factor score - Uncontrolled Hostility/Excitement Score for participants was calculated as the sum of the rating assigned to each of the 4 items, and ranged from 4 to 28 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Brexpiprazole 4mg: Brexpiprazole 4mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of placebo over a 1-week period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose the day after the Week 1 visit (ie, the beginning of Week 2).
- Brexpiprazole 2mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of placebo over a 5-day period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose by Day 5.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 123 | 56 | 108
Units on a scale | -1.90 (0.28) | -1.91 (0.28) | -1.15 (0.41) | -0.82 (0.30)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.0085, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.07, 95% CI 2-sided [-1.87 to -0.28]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0081, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -1.08, 95% CI 2-sided [-1.88 to -0.28]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.5172, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -0.33, 95% CI 2-sided [-1.31 to 0.66]

16. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Anxiety Depression Score
Description: The PANSS Marder Factor score - Anxiety/Depression Score consists of 4 PANSS items (anxiety [G2], guilt feelings [G3], tension [G4], depression [G6]). The PANSS Marder Factor score - Anxiety/Depression Score for participants was calculated as the sum of the rating assigned to each of the 4 items, and ranged from 4 to 28 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2mg | Brexpiprazole 0.25mg | Placebo
Number analyzed (Participants) | 121 | 123 | 56 | 108
Units on a scale | -3.40 (0.25) | -3.70 (0.25) | -3.27 (0.35) | -3.05 (0.26)
Statistical Analysis 1: Comparison: Brexpiprazole 4mg vs Placebo; Test type: Superiority or Other; p = 0.3284, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -0.34, 95% CI 2-sided [-1.03 to 0.35]
Statistical Analysis 2: Comparison: Brexpiprazole 2mg vs Placebo; Test type: Superiority or Other; p = 0.0655, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -0.65, 95% CI 2-sided [-1.34 to 0.04]
Statistical Analysis 3: Comparison: Brexpiprazole 0.25mg vs Placebo; Test type: Superiority or Other; p = 0.6251, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; Treatment difference = -0.21, 95% CI 2-sided [-1.07 to 0.64]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time the participant signs the informed consent form, throughout the 6-week treatment period and until 30 days after the last dose of study medication.
Groups:
- Brexpiprazole 2 mg: Brexpiprazole 2mg tablet once daily for 6 weeks.
  Participants were titrated to the target dose of brexpiprazole over a 5-day period beginning at the randomization (Day 1), and all participants were to have achieved the assigned dose by Day 5.
- Brexpiprazile 0.25 mg: Brexpiprazole 0.25mg tablet once daily for 6 weeks.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 2 mg | Brexpiprazile 0.25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/180 | 4/182 | 4/90 | 7/184
Other Adverse Events (participants affected / at risk) | 64/180 | 53/182 | 25/90 | 65/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 4mg (N=180) | Brexpiprazole 2 mg (N=182) | Brexpiprazile 0.25 mg (N=90) | Placebo (N=184)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 1 | 2
Schizophrenia (Psychiatric disorders) | 2 | 2 | 2 | 2
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 4mg (N=180) | Brexpiprazole 2 mg (N=182) | Brexpiprazile 0.25 mg (N=90) | Placebo (N=184)
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 5 | 3
Nausea (Gastrointestinal disorders) | 6 | 10 | 1 | 8
Akathisia (Nervous system disorders) | 13 | 8 | 0 | 4
Headache (Nervous system disorders) | 22 | 17 | 9 | 15
Agitation (Psychiatric disorders) | 13 | 11 | 4 | 19
Insomnia (Psychiatric disorders) | 15 | 16 | 8 | 18
Schizophrenia (Psychiatric disorders) | 10 | 7 | 6 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No